CLINICAL TRIAL: NCT02954380
Title: The Comparative Efficacy of the Zio Patch vs Implantable Loop Recorder in Atrial Fibrillation
Acronym: ALERT-AF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ir-iis-01 JAX
Record Dates: First submitted 2016-11-01; First posted 2016-11-03 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ZIO/ILR (Experimental): THe Zio ILR arm will already have an ILR implanted for standard of care and will receive the Zio patch
  Interventions: Device: Zio

INTERVENTIONS:
Device: Zio — long term continuous monitoring

SUMMARY:
The aim of our study is to investigate if LTCM's are superior to implantable loop recorders in detecting atrial fibrillation after pulmonary vein isolation. This study will provide insights on a possible alternative for detection of arrhythmia.

DETAILED DESCRIPTION:
Summary Atrial fibrillation (AF) is the most common arrhythmia, increasing in prevalence with age characterized by chaotic contraction of the atrium. An estimated 2.2 million people in the United States and 4.5 million in the European Union have AF.[1,2] AF is associated with heart failure, hemodynamic impairment, and symptoms affecting quality of life. Patients have an increased risk of thromboembolic events, including stroke, resulting in significant morbidity, mortality, and costs. [1-5]

Diagnosis of atrial fibrillation is made via an electrocardiogram (ECG) recording. Any arrhythmia that has the ECG characteristics of AF and lasts sufficiently long for a 12-lead ECG to be recorded, or at least 30 seconds on a rhythm strip, should be considered an AF episode.[6] The diagnosis requires an ECG or rhythm strip demonstrating: 1) "absolutely" irregular RR intervals (in the absence of complete AV block), 2) Absence of distinct P waves on the surface ECG, and 3) an atrial cycle length (when visible) that is usually variable and less than 200 msec. [7]

During the past decade, catheter ablation of atrial fibrillation (AF) has evolved rapidly from an investigational procedure to its current status as a commonly performed ablation procedure in many major hospitals throughout the world. The goal of the ablation is to isolate the pulmonary veins from which in the majority of the population atrial fibrillation originates. During the past several years a large number of meta analyses have been performed in the hope of better defining the efficacy of AF ablation. Overall, the success rate was 77.8% in the ablation arm as compared with 23.3% in the control group.

Catheter ablation has decreased the recurrence of AF by 71% (relative risk 0.29). Several other meta analyses of randomized clinical trials have confirmed these findings [8-12].

Background and Significance Arrhythmia monitoring in patients undergoing atrial fibrillation ablation is challenging. Trans-telephonic monitors (TTMs) are cumbersome to use and provide limited, temporal assessment. Implantable loop recorders may overcome these limitations. The ABACUS study sought to evaluate the utility of implantable loop recorders (ILRs) versus conventional monitoring (CM) in patients undergoing AF ablation. In AF ablation patients, ILR detected more arrhythmias than CM. However, false detection remained a challenge including the inability to the ILR to detect atrial fibrillation less than 2 minutes in duration. The investigators concluded that with adequate oversight, ILRs may be useful in monitoring these patients after ablation. [13] ILR's have been convenient to patients due to the fact that they do not require electrodes or patches. In addition there is no external monitor that must be accompanied with the electrode adhesive pair.

Despite the convenience of the ILR with respect to everyday life, there is an offset to diagnostic sensitivity given inherent algorithms limiting the fastest time to detection 2 minutes. Current Heart Rhythm Consensus 2012 HRS/EHRA/ECAS Expert Consensus Statement on Catheter and Surgical Ablation of Atrial Fibrillation: Recommendations for Patient Selection, Procedural Techniques, Patient Management and Follow-up, Definitions, Endpoints, and Research Trial DesignS consensus demonstrates 30 seconds as deemed clinically acceptable for duration of atrial fibrillation. Despite advances in technology patients can frequently experience recurrence of atrial fibrillation either after cardioversion or post atrial fibrillation ablation.

Implantable loop recorders have emerged as a technology which requires a surgical procedure and can potentially record continuous rhythm for its battery life which usually lasts approximately three years. The procedure can also lead to explantation secondary to erosion or migration. Some cardiologists and electrophysiologists use the ILR post ablation for AF surveillance. This affords long term surveillance, however the device is costly and there is a risk of infection as well. Novel technology termed LTCM has the capability to record and store continuous ECG for up to 14 days.

Novel technology available termed ambulatory long term continuous monitor (LTCM) one of which includes Zio XT has the capability to record and store continuous ECG for up to 14 days. Long Term Cardiac Telemetry provides beat-to-beat ECG recording, storage and analysis with automatic arrhythmia detection. The ZIO XT device utilizes an adhesive patch which attaches conveniently to the patient. The LTCM has the capability to detect AF of duration less than 2 minutes when compared to the ILR. The patches are disposable and may be worn for up to 14 days duration. . The Zio patch They contains a proprietary algorithm which can detect a number of different arrhythmias including but not limited to non-sustained ventricular tachycardia, brady- arrhythmia including heart block as well as life threatening polymorphic ventricular tachycardia. LTCMs are substantially cost effective and may be used in clinics or emergency departments. The LTCMs however have not been studied in a comparative effectiveness trial with implantable loop recorders.

Each patient will already have an implantable loop recorder and will receive the Zio patch as the experimental arm of the trial.

The primary endpoint of our investigation is to compare LTCM's verses implantable loop recorders in successful detection and recurrence of atrial fibrillation after pulmonary vein isolation. We hypothesize the LTCM's will detect atrial fibrillation after pulmonary vein isolation more accurately than the implantable loop recorders. Secondary objectives will be the comparisons of the following:

1. Agreement between the assessment of events between the two devices.
2. Sensitivity, Specificity, PPV, Accuracy and Reliability of each of the two devices of (LTCM vs. ILR) compared to the ECG readout of each. That is, the ECG from the LCTM will be used as the gold standard to assess the LCTM events and the ECG from the ILR will be used to assess the ILR events. Summary statistics from these two events will be presented side by side.
3. Successful symptom rhythm correlation judged by using a patient activator on the patch
4. Signal Quality in Voltage of ILR vs. LTCM
5. Rate of False Detection in ILR vs. LTCM
6. Quality of Monitoring Experience Survey of the patient
7. Cost Benefit Analysis

7. Economic outcomes 8. Arrhythmia other than AF detected

Research Plan Inclusion Criterion

1. Patients with a diagnosis of paroxysmal or persistent atrial fibrillation documented on electrocardiography
2. Patients must already have a Medtronic LINQ ILR as standard of care already implanted as standard of care
3. Patients must be available for at least 7 but maximum of 14 days after patch application
4. Patients must be greater than or equal to 18 years old.

Exclusion Criterion

Patients less than 18 years of age

1. Patients with a history of permanent atrial fibrillation
2. Patients with an implanted pacemaker or implantable cardioverter defibrillator
3. CPatients with cognitive delay and or dementia
4. UPatients unable to give Consent.
5. Patients with adhesive allergy

Research Design The study will be performed at the University of Florida Health Science Center at UF Health, Jacksonville-Division of Cardiology. Patients will be recruited in the Cardiology Clinics of our institution and will be screened by Cardiology Research Staff, who will verify all candidates meet inclusion and exclusion criteria.

Patients found eligible for this study will already have undergone an implantable loop recorder (ILR) (Medtronic LINQ, Minneapolis, MN) implant. After providing written informed consent, subjects will be paired with a LTCM - ZIO® Patch, iRhythm Technologies, Inc. San Francisco, CA).

Both the ILR and ZIO Patch will be set to Eastern Standard Time (EST). Subjects will be instructed to wear the ZIO Patch for a minimum of 7 days but not exceeding 14 days.

To help ensure compliance a study follow up phone call will be made at day 7 (+/- 1 day).

Subjects will return to UF Shands -Jacksonville on day 12 (+/- 2 days) for removal of the patch and data download of ILR. Quality of Monitoring Questionnaire will be provided.

To avoid reporting bias raw data from the ZIO Patch, raw data of the event recording (ECG analysis)will be reviewed by an adjudication committee of two three board certified cardiologists. If there is disagreement, a third physician will decide.

At the final study visit (as outlined in METHODS) the patch will be shipped to iRhythm.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of paroxysmal or persistent atrial fibrillation documented on electrocardiography
2. Patients must already have a Medtronic LINQ ILR as standard of care already implanted as standard of care
3. Patients must be available for at least 7 but maximum of 14 days after patch application
4. Patients must be greater than or equal to 18 years old.

Exclusion Criteria:

1. Patients with a history of permanent atrial fibrillation
2. Patients with an implanted pacemaker or implantable cardioverter defibrillator
3. Patients with cognitive delay and or dementia
4. Patients unable to give Consent.
5. Patients with adhesive allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Agreement between the assessment of events between the two devices | 10 days

SECONDARY OUTCOMES:
Sensitivity, Specificity, PPV, Accuracy and Reliability | 10 days
  the ECG from the LCTM will be used as the gold standard to assess the LCTM events and the ECG from the ILR will be used to assess the ILR events.
Signal quality | 10 days
  Measured in Voltage from baseline

CONTACTS AND LOCATIONS:
Overall Officials: John N Catanzaro, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fuster V, Ryden LE, Cannom DS, Crijns HJ, Curtis AB, Ellenbogen KA, Halperin JL, Le Heuzey JY, Kay GN, Lowe JE, Olsson SB, Prystowsky EN, Tamargo JL, Wann S, Smith SC Jr, Jacobs AK, Adams CD, Anderson JL, Antman EM, Halperin JL, Hunt SA, Nishimura R, Ornato JP, Page RL, Riegel B, Priori SG, Blanc JJ, Budaj A, Camm AJ, Dean V, Deckers JW, Despres C, Dickstein K, Lekakis J, McGregor K, Metra M, Morais J, Osterspey A, Tamargo JL, Zamorano JL; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; European Society of Cardiology Committee for Practice Guidelines; European Heart Rhythm Association; Heart Rhythm Society. ACC/AHA/ESC 2006 Guidelines for the Management of Patients with Atrial Fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the European Society of Cardiology Committee for Practice Guidelines (Writing Committee to Revise the 2001 Guidelines for the Management of Patients With Atrial Fibrillation): developed in collaboration with the European Heart Rhythm Association and the Heart Rhythm Society. Circulation. 2006 Aug 15;114(7):e257-354. doi: 10.1161/CIRCULATIONAHA.106.177292. No abstract available. PMID 16908781
- [Background] Chugh SS, Blackshear JL, Shen WK, Hammill SC, Gersh BJ. Epidemiology and natural history of atrial fibrillation: clinical implications. J Am Coll Cardiol. 2001 Feb;37(2):371-8. doi: 10.1016/s0735-1097(00)01107-4. PMID 11216949
- [Background] Flaker GC, Belew K, Beckman K, Vidaillet H, Kron J, Safford R, Mickel M, Barrell P; AFFIRM Investigators. Asymptomatic atrial fibrillation: demographic features and prognostic information from the Atrial Fibrillation Follow-up Investigation of Rhythm Management (AFFIRM) study. Am Heart J. 2005 Apr;149(4):657-63. doi: 10.1016/j.ahj.2004.06.032. PMID 15990749
- [Background] Glotzer TV, Hellkamp AS, Zimmerman J, Sweeney MO, Yee R, Marinchak R, Cook J, Paraschos A, Love J, Radoslovich G, Lee KL, Lamas GA; MOST Investigators. Atrial high rate episodes detected by pacemaker diagnostics predict death and stroke: report of the Atrial Diagnostics Ancillary Study of the MOde Selection Trial (MOST). Circulation. 2003 Apr 1;107(12):1614-9. doi: 10.1161/01.CIR.0000057981.70380.45. Epub 2003 Mar 24. PMID 12668495
- [Background] Capucci A, Santini M, Padeletti L, Gulizia M, Botto G, Boriani G, Ricci R, Favale S, Zolezzi F, Di Belardino N, Molon G, Drago F, Villani GQ, Mazzini E, Vimercati M, Grammatico A; Italian AT500 Registry Investigators. Monitored atrial fibrillation duration predicts arterial embolic events in patients suffering from bradycardia and atrial fibrillation implanted with antitachycardia pacemakers. J Am Coll Cardiol. 2005 Nov 15;46(10):1913-20. doi: 10.1016/j.jacc.2005.07.044. Epub 2005 Oct 24. PMID 16286180
- [Background] Calkins H, Brugada J, Packer DL, Cappato R, Chen SA, Crijns HJ, Damiano RJ Jr, Davies DW, Haines DE, Haissaguerre M, Iesaka Y, Jackman W, Jais P, Kottkamp H, Kuck KH, Lindsay BD, Marchlinski FE, McCarthy PM, Mont JL, Morady F, Nademanee K, Natale A, Pappone C, Prystowsky E, Raviele A, Ruskin JN, Shemin RJ; Heart Rhythm Society; European Heart Rhythm Association; European Cardiac Arrhythmia Society; American College of Cardiology; American Heart Association; Society of Thoracic Surgeons. HRS/EHRA/ECAS expert consensus statement on catheter and surgical ablation of atrial fibrillation: recommendations for personnel, policy, procedures and follow-up. A report of the Heart Rhythm Society (HRS) Task Force on Catheter and Surgical Ablation of Atrial Fibrillation developed in partnership with the European Heart Rhythm Association (EHRA) and the European Cardiac Arrhythmia Society (ECAS); in collaboration with the American College of Cardiology (ACC), American Heart Association (AHA), and the Society of Thoracic Surgeons (STS). Endorsed and approved by the governing bodies of the American College of Cardiology, the American Heart Association, the European Cardiac Arrhythmia Society, the European Heart Rhythm Association, the Society of Thoracic Surgeons, and the Heart Rhythm Society. Europace. 2007 Jun;9(6):335-79. doi: 10.1093/europace/eum120. No abstract available. PMID 17599941
- [Background] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Popescu BA, Schotten U, Van Putte B, Vardas P, Agewall S, Camm J, Baron Esquivias G, Budts W, Carerj S, Casselman F, Coca A, De Caterina R, Deftereos S, Dobrev D, Ferro JM, Filippatos G, Fitzsimons D, Gorenek B, Guenoun M, Hohnloser SH, Kolh P, Lip GY, Manolis A, McMurray J, Ponikowski P, Rosenhek R, Ruschitzka F, Savelieva I, Sharma S, Suwalski P, Tamargo JL, Taylor CJ, Van Gelder IC, Voors AA, Windecker S, Zamorano JL, Zeppenfeld K. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Eur J Cardiothorac Surg. 2016 Nov;50(5):e1-e88. doi: 10.1093/ejcts/ezw313. Epub 2016 Sep 23. No abstract available. PMID 27663299
- [Background] Noheria A, Kumar A, Wylie JV Jr, Josephson ME. Catheter ablation vs antiarrhythmic drug therapy for atrial fibrillation: a systematic review. Arch Intern Med. 2008 Mar 24;168(6):581-6. doi: 10.1001/archinte.168.6.581. PMID 18362249
- [Background] Nair GM, Nery PB, Diwakaramenon S, Healey JS, Connolly SJ, Morillo CA. A systematic review of randomized trials comparing radiofrequency ablation with antiarrhythmic medications in patients with atrial fibrillation. J Cardiovasc Electrophysiol. 2009 Feb;20(2):138-44. doi: 10.1111/j.1540-8167.2008.01285.x. Epub 2008 Sep 3. PMID 18775040
- [Background] Parkash R, Tang AS, Sapp JL, Wells G. Approach to the catheter ablation technique of paroxysmal and persistent atrial fibrillation: a meta-analysis of the randomized controlled trials. J Cardiovasc Electrophysiol. 2011 Jul;22(7):729-38. doi: 10.1111/j.1540-8167.2011.02010.x. Epub 2011 Feb 18. PMID 21332861
- [Background] Piccini JP, Lopes RD, Kong MH, Hasselblad V, Jackson K, Al-Khatib SM. Pulmonary vein isolation for the maintenance of sinus rhythm in patients with atrial fibrillation: a meta-analysis of randomized, controlled trials. Circ Arrhythm Electrophysiol. 2009 Dec;2(6):626-33. doi: 10.1161/CIRCEP.109.856633. PMID 20009077
- [Background] Kapa S, Epstein AE, Callans DJ, Garcia FC, Lin D, Bala R, Riley MP, Hutchinson MD, Gerstenfeld EP, Tzou W, Marchlinski FE, Frankel DS, Cooper JM, Supple G, Deo R, Verdino RJ, Patel VV, Dixit S. Assessing arrhythmia burden after catheter ablation of atrial fibrillation using an implantable loop recorder: the ABACUS study. J Cardiovasc Electrophysiol. 2013 Aug;24(8):875-81. doi: 10.1111/jce.12141. Epub 2013 Apr 11. PMID 23577826